CLINICAL TRIAL: NCT01212380
Title: A Phase I Study of Carfilzomib in Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL)/Prolymphocytic Leukemia (PLL)
Brief Title: Study of Carfilzomib in Chronic Lymphocytic Leukemia (CLL), Small Lymphocytic Lymphoma (SLL) or Prolymphocytic Leukemia (PLL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Jennifer Woyach, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-09108; NCI-2010-01884 (Registry Identifier: CTRP (Clinical Trial Registration Program))
Record Dates: First submitted 2010-09-10; First posted 2010-09-30 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Hematopoietic/Lymphoid Cancer; Prolymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Prolymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Hematologic Neoplasms; Leukemia, Prolymphocytic | interventions — carfilzomib; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Patients receive carfilzomib IV over 30 minutes once daily on days 1, 2, 8, 9, 15, and 16. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.Performance of pharmacology, pharmacodynamic and pharmacogenomic studies allow assessment of carfilzomib mechanism of action and also to understand how the variability of these different features correlate with clinical benefit/response and also toxicity.
  Interventions: Drug: carfilzomib; Other: Cytokine Assessment; Other: Pharmacodynamic Studies; Other: Proteosome Inhibition Assessment; Other: Pharmacogenomic Studies

INTERVENTIONS:
Drug: carfilzomib — Given IV infusion lasting 30 minutes. Will be administered IV at a specified dose in mg/m2 QDx2 weekly for 3 weeks (days 1, 2, 8, 9, 15, and 16). The first and second dose will always be administered at 20 mg/m2.
  Other Names: PR-171
Other: Cytokine Assessment — TNF-α,IFN-γ,IL-6,IL-8,IL-10,and IL-1β pre-dose, completion, 30 minutes, 2 hours, 6 hours, and approximately 24 hours from initiation of therapy on days 1 and 8 of treatment. These will be assessed utilizing standard ELISA or flow cytometry methodology. Other cytokines or soluble factors may be assessed that relate to drug toxicity or response. After 6 patients are examined in each group, the time points or number of cytokines examined may be changed to decrease time points examined. Cytokines will be examined by a multiplex flow cytometry assay or ELISA. Other cytokines, chemokines, or soluble factors may be assessed on residual material not used for these studies.
  Other Names: correlative studies
Other: Pharmacodynamic Studies — Based upon our preliminary data changes occuring in vivo during carfilzomib treatment will be determined and if their occurrence correlates with both clinical response and development of cytokine release. These studies will be performed from CD19 selected CLL cells at screening, pre-treatment, 4 hours, and 24 hours post-therapy on days 1 and 8 of treatment; end of therapy evaluation, and at time of relapse (in responding patients). These studies will include assessment of NF-κB (p50/p65 binding; I-κB level, P-I-κB level, select target genes), p53 (p53 nuclear levels, p53 nuclear binding, and select target genes), p73, and ER stress response. Standard Western Blot, EMSA, RT-PCR will be done to complete these studies.
  Other Names: correlative studies
Other: Proteosome Inhibition Assessment — Proteosome inhibition on CLL cells will be examined at screening, pre-treatment and post-treatment (immediately after completion of drug) days 1, pre-treatment day 2, day 3 (optional), day 5 (optional),pre and post-treatment days 8, pre and post-treatment days 9, day 10 (optional),day 12 (optional), and day 15 (optional).
  Other Names: pharmacological studies
Other: Pharmacogenomic Studies — Germ line DNA from a buccal swab and bone marrow fibroblasts will be obtained at baseline screening for possible examination of SNP polymorphisms that may correlate with response and toxicity to carfilzomib therapy. Tumor DNA will be derived from samples obtained at baseline for the p53 mutational studies. SNPs related to drug metabolism, response, or toxicity to therapy, cytokine release, and tumor biology may be examined. Other SNPs may be used in the future. Given the potential for contamination in the recipient, recipient DNA from a buccal swab and/or saliva will be obtained at baseline screening for examination of SNP polymorphisms that may correlate with response, toxicity, and pharmacokinetics.
  Other Names: correlative studies

SUMMARY:
RATIONALE:

Carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE:

This phase I trial is studying the side effects and the best dose of carfilzomib in treating patients with relapsed or refractory chronic lymphocytic leukemia(CLL),small lymphocytic lymphoma(SLL), or prolymphocytic leukemia (PLL).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dose limiting toxicity (DLT) and maximal tolerated dose (MTD) of carfilzomib in patients with relapsed or refractory Chronic Lymphocytic Leukemia(CLL) / Small Lymphocytic Lymphoma (SLL) and Prolymphocytic Leukemia (PLL).

II. To evaluate the safety and toxicity profile of carfilzomib in relapsed or refractory chronic lymphocytic leukemia (CLL)/small lymphocytic leukemia (SLL)/prolymphocytic leukemia (PLL).

SECONDARY OBJECTIVES:

I. To evaluate efficacy of carfilzomib therapy in relapsed or refractory chronic lymphocytic leukemia (CLL)/small lymphocytic leukemia (SLL)/prolymphocytic leukemia (PLL) to justify future phase II studies.

II. To determine the degree and duration of cellular proteosome inhibition induced by carfilzomib and relationship of this to pharmacodynamics, response and toxicity.

III. To determine the pharmacokinetics (plasma and cellular) of carfilzomib and relationship of this to proteosome inhibition, pharmacodynamics, response, and toxicity.IV. To examine the effect of carfilzomib on pharmacodynamic parameters including cytokines, changes in downstream targets including NF-kappa B (p50/p65 binding; I-kappa B level, P-I-kappa B level,select target genes), p53 (p53 nuclear levels, p53 nuclear binding, and select target genes), ER stress proteins, and p73.

OUTLINE: This is a dose-escalation study of carfilzomib.Patients receiving carfilzomib intra-venous(IV) over 30 minutes once daily, on days 1, 2, 8, 9, 15, and 16. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated patients with a diagnosis of chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma (SLL), or prolymphocytic leukemia (PLL) by NCI Criteria with intermediate or high risk B-Cell chronic lymphocytic leukemia (CLL)(Modified Rai stage) satisfying at least one of the criteria for active disease requiring treatment;patients with a history of Richter's transformation are eligible if they now have evidence of chronic lymphocytic leukemia (CLL) only, with < 10% large cells in the bone marrow
* Massive or progressive splenomegaly and/or lymphadenopathy; or need for cytoreduction for stem cell transplant
* Anemia (hemoglobin < 11 g/dl) or thrombocytopenia (platelets < 100 x 10^9/L)
* Presence of weight loss > 10% over the preceding 6 month period
* NCI grade 2 or 3 fatigue
* Fevers > 100.5 °C or night sweats for greater than 2 weeks without evidence of infection
* Progressive lymphocytosis with an increase of > 50% over a 2 month period or an anticipated doubling time of less than 6 months
* Creatinine Clearance (CrCl) > 15mL/min
* Alanine aminotransferase (ALT) < 3X upper limit of normal (ULN)
* Bilirubin =< 2 times the upper limit of normal, unless disease related
* Platelets >= 20 x 10^9/L and absence of active bleeding
* Patients must have an ECOG (Eastern Cooperative Oncology Group) performance status =< 2
* Patients must not have secondary cancers that result in a life expectancy of <2 years or that would confound assessment of toxicity in this study
* Patients of all racial/ethnic groups are eligible for the study if they meet eligibility criteria outlined-
* Patients must provide written informed consent

Exclusion Criteria:

* Absence of previously treated chronic lymphocytic leukemia (CLL)
* Female subject that is pregnant or breastfeeding; women of childbearing potential and men must agree to use adequate contraception prior to study entry, duration of study participation,and 30 days following study completion; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately;confirmation that the subject is not pregnant must be established by a negative serum -human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening; pregnancy testing is not required for post-menopausal or surgically sterilized women
* Patients with congestive heart failure (CHF)in whom pre-treatment hydration would be prohibitive;New York Heart Association (NYHA) Class III/IV CHF is excluded
* Patients who have had treatment for chronic lymphocytic leukemia (CLL) within 2 weeks, although palliative steroids are acceptable
* Patient unable to give written informed consent
* Failure to recover from toxicity of previous radiotherapy or chemotherapy to grade 1
* Patients with active infections requiring intravenous (IV) antibiotic/antiviral therapy are not eligible for entry onto the study until resolution of the infection; patients on prophylactic antibiotics or antivirals are acceptable
* Patients who have previously taken bortezomib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-10; Primary Completion 2014-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Determine safety of carfilzomib by evaluating the toxicity profile. | Up to 24 months
  The safe use of carfilzomib will be assessed by:
  * Determining the dose limiting toxicity and maximal tolerated dose of carfilzomib in patients with relapsed or refractory chronic lymphocytic leukemia (CLL)/small lymphocytic leukemia (SLL) and prolymphocytic leukemia (PLL)
  * To evaluating the toxicity profile of carfilzomib in relapsed or refractory chronic lymphocytic leukemia (CLL)/small lymphocytic leukemia (SLL) and prolymphocytic leukemia (PLL)

SECONDARY OUTCOMES:
To evaluate the efficacy of Carfilzomib therapy in relapsed or refractory chromic lymphocytic leukemia (CLL)/small lymphocytic leukemia (SLL)/prolymphocytic leukemia (PLL) | Up to 24 months
  Efficacy of this therapy is evaluated by:
  * Determining the degree and duration of cellular proteosome inhibition and relationship to pharmacodynamic (PD), response and toxicity.
  * Determining the pharmacokinetics(plasma and cellular)of carfilzomib and relationship to proteosome inhibition, PD, response and toxicity.
  * Examining the effect of carfilzomib on PD parameters, changes in downstream targets including NFkB (p50/p65 binding;IkB level, P-IkB level, select target genes), p53 (p53 nuclear levels, p53 nuclear binding, and select target genes), ER stress proteins, and p73

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Woyach, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu